CLINICAL TRIAL: NCT04729218
Title: The Movement Imagery Ability in Patients With Familial Mediterranean Fever
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Albina Alikaj, Principal Investigator, Medipol University
Other Study IDs: 10840098-604.01.01-E.399988
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Familial Mediterranean Fever
Keywords: movement imagery ability; pain; catastrophizing; familial mediterranean fever
MeSH Terms: conditions — Familial Mediterranean Fever; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Familial Mediterranean Fever group: 30 participants
  Interventions: Behavioral: movement imagery ability
- Healthy group: 30 participants
  Interventions: Behavioral: movement imagery ability

INTERVENTIONS:
Behavioral: movement imagery ability — Determining the movement imagery ability: internal visual, external visual and kinesthetic imagery

SUMMARY:
Motor imagery is the mental representation of movement without any doing body movement. A main function of imagery is to aid the self-regulation of thoughts, feelings, and behaviours. Studies have shown to be more effective for individuals displaying a higher level of imagery ability when using imagery to improve motor and motivational outcomes, including self-efficacy. The aim of this study is to measure the movement imagery ability in patients with Familial Mediterranean Fever and compare it with healthy individuals.

DETAILED DESCRIPTION:
Familial Mediterranean Fever (FMF) is an autosomal recessive disease characterized by recurrent and self-limited attacks of fever associated with abdominal, chest, and joint pain. Previous studies have shown that individuals with FMF are more limited in terms of physical function than the normal population, and depression and anxiety are more common in these individuals. Being a lifetime disease, quality of life, and mental health can be affected due to serious complications such as attack frequency, disease resistance, and sometimes amyloidosis. Mental imagery is the ability to imaging the movement without doing the physical execution of the movement. During the last years, mental imagery is used in clinical practice as a tool for the treatment of chronic pain. Pain differs in patients with rheumatic diseases. Stress is one of the predictors of pain in patients with FMF. Even if the frequency is variable when attacks happen they may affect patients physically and their mental health and the ability to cope. A main function of imagery is to aid the self-regulation of thoughts, feelings, and behaviors. To use imagery for motor and motivational outcomes firstly the imagery ability levels should be measured.

ELIGIBILITY:
Inclusion Criteria:

* having had at least one attack last year
* co-operated individuals

Exclusion Criteria:

* patients with a neurological disorder,
* diagnosed with cancer,
* cognitive impairment,
* having a primary pathology of the musculoskeletal system,
* having previous imagery practice,
* having an additional rheumatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Familial Mediterranean Fever and Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Movement Imagery Questionnaire-3 (MIQ-3) | Baseline
  It is a questionnaire containing 12 items to evaluate the visual imagination skills of the individual. It evaluates internal visual imagery, external visual imagery, and kinesthetic imagery. For each item, first of all, individuals read the description of the movement, and then it is desired to perform the movement physically and after that, the same movement is requested. Individuals evaluate the degree of imagination on a 7-point Likert-type scale ranging from 1 (very difficult to see/feel) to 7 (very easy to see/feel). The motion visualization questionnaire has good psychometric properties, internal reliability, and estimated validity.

SECONDARY OUTCOMES:
McGill Melzack Pain Questionnaire (MPQ) | Baseline
  MPQ consists of 78 descriptors grouped into four categories: sensory, affective, evaluative, and miscellaneous. These four categories were grouped into 20 subclasses each made up of 2 to 6 words according to pain intensity. Patients were asked to choose the pain descriptors according to the type of pain they felt during the attack episodes. Patients were instructed to choose one of the words that best described their type of pain experience. Changing of pain with time was assessed. Pain right now, pain at its worst and pain at its least was evaluated. Pain exacerbating or relieving factors were recorded.
Pain Catastrophizing Scale | Baseline
  Pain Catastrophizing Scale identifies catastrophic thoughts or feelings and ineffective coping strategies of patients. PCS is a Likert-type self-assessment scale consisting of thirteen items. Each item is evaluated between 0 and 4 points. The total score ranges from 0 to 52. Includes rumination, magnification, and helplessness subscales. High scores indicate that the level of disaster is high.

CONTACTS AND LOCATIONS:
Overall Officials: Albina Alikaj, MSc, Principal Investigator — Medipol University; Ahsen Büyükaslan, MSc, Study Chair — Medipol University; Serdal Uğurlu, Prof, Study Director — Istanbul University - Cerrahpasa; Burcu Dilek, PhD, Study Director — Acibadem University
Locations (1):
- Istanbul University, Cerrahpaşa Medical Faculty, Department of Rheumatology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Reliability and validity of the Turkish version of the movement imagery questionnaire-3: Its cultural adaptation and psychometric properties — http://www.nsnjournal.org/article.asp?issn=2636-865X;year=2020;volume=37;issue=4;spage=221;epage=227;aulast=Dilek